CLINICAL TRIAL: NCT01530035
Title: Cardiovascular and Muscular Adaptations to Recreational Soccer and Strength Training in Elderly Healthy 65-75-year-old Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jakob Friis Schmidt, MD PhD student, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-1-2011-013
Record Dates: First submitted 2012-01-26; First posted 2012-02-09 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Adaptation Reaction
Keywords: cardiac; vascular; muscular; adaptations; soccer training; strength training
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- soccer training intervention (Active Comparator)
  Interventions: Other: physical training
- strength training intervention (Other)
  Interventions: Other: physical training
- control group (No Intervention): elderly men with no change in daily activities
- active soccer control group (No Intervention): veteran soccer players with a 40 year history of continues soccer playing

INTERVENTIONS:
Other: physical training — training
  Arms: soccer training intervention; strength training intervention

SUMMARY:
A one-year intervention study of 41 healthy elderly men aged 65-75-years.Of these, 24 subjects are untrained men with no regular training activity for the last 5 years. After medical screening and pre-testing, they will be randomized into a football group (n=9), a strength-training group (n=9) or a sedentary control group (n=6). Additional 17 subjects are recruited from local football clubs and have been active football players for the last 40 years. Training will be performed 3x1 hour per week and evaluation will take place after 0, 3 and 12 months. Primary endpoints will be changes in cardiac and vascular structure and function measured by advanced echocardiography (tissue Doppler and speckle tracking imaging), and peripheral arterial tonometry (Endo---PAT device). Secondary endpoints will be evaluation of potential changes in VO2 max, blood pressure, muscle capillaries, lipid profile, circulating catecholamines, body composition, and insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* 65-75 year old men
* healthy
* non-smoking
* non-hypertension
* non- cardiac disease

Exclusion Criteria:

* smoking
* cardiac disease
* biomechanical disorders
* cardiac medication

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
cardiac adaptations | after 16 weeks and one year
  changes in cardiac function after 16 weeks and one year measured by advanced echocardiography (tissue Doppler and speckle tracking imaging)

SECONDARY OUTCOMES:
Cardiorespiratory fitness, muscular adaptations, Bloodpressure and Glucose tolerance | after 16 weeks and one year
  Improvements in cardiorespiratory fitness assessed with VO2 max treadmill testing.
  Changes in muscular tissue with biopsies from the vastus lateralis muscle. Changes in resting blood pressure in incline postion Changes in glucose tolerance with oral glucose tolerance testing

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bangsbo, professor, Study Chair — Institute of exercise and sports sciences, university of copenhagen Denmark
Locations (1):
- Institute of exercise and sports sciences, university of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen TR, Schmidt JF, Pedersen MT, Krustrup P, Bangsbo J. The Effects of 52 Weeks of Soccer or Resistance Training on Body Composition and Muscle Function in +65-Year-Old Healthy Males--A Randomized Controlled Trial. PLoS One. 2016 Feb 17;11(2):e0148236. doi: 10.1371/journal.pone.0148236. eCollection 2016. PMID 26886262
- [Derived] Andersen TR, Schmidt JF, Nielsen JJ, Randers MB, Sundstrup E, Jakobsen MD, Andersen LL, Suetta C, Aagaard P, Bangsbo J, Krustrup P. Effect of football or strength training on functional ability and physical performance in untrained old men. Scand J Med Sci Sports. 2014 Aug;24 Suppl 1:76-85. doi: 10.1111/sms.12245. Epub 2014 Jun 5. PMID 24903323
- [Derived] Helge EW, Andersen TR, Schmidt JF, Jorgensen NR, Hornstrup T, Krustrup P, Bangsbo J. Recreational football improves bone mineral density and bone turnover marker profile in elderly men. Scand J Med Sci Sports. 2014 Aug;24 Suppl 1:98-104. doi: 10.1111/sms.12239. Epub 2014 Jun 5. PMID 24903207
- [Derived] Schmidt JF, Hansen PR, Andersen TR, Andersen LJ, Hornstrup T, Krustrup P, Bangsbo J. Cardiovascular adaptations to 4 and 12 months of football or strength training in 65- to 75-year-old untrained men. Scand J Med Sci Sports. 2014 Aug;24 Suppl 1:86-97. doi: 10.1111/sms.12217. Epub 2014 Jun 5. PMID 24902992